CLINICAL TRIAL: NCT04192435
Title: Tranexamic Acid to Reduce Infection After Gastrointestinal Surgery; The TRIGS Trial
Brief Title: Tranexamic Acid to Reduce Infection After Gastrointestinal Surgery
Acronym: TRIGS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 087
Record Dates: First submitted 2019-11-27; First posted 2019-12-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Infection Wound; Gastrointestinal Complication; Anesthesia; Bleeding; Healthcare Associated Infection
MeSH Terms: conditions — Wound Infection; Hemorrhage; Cross Infection | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, randomised trial of TxA versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matched TxA and placebo vials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): At induction of anesthesia and prior to surgical incision a bolus of 0.15 ml/kg ( up to a maximum of 15 ml) , and then commence an infusion of 0.05 ml/kg/h until the end of surgery. The total maximal administered study drug volume will be 30 ml.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): At induction of anesthesia and prior to surgical incision a bolus of 0.15 ml/kg ( up to a maximum of 15 ml) , and then commence an infusion of 0.05 ml/kg/h until the end of surgery. The total maximal administered study drug volume will be 30 ml.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tranexamic Acid — 100mg/ml
  Arms: Tranexamic acid
Drug: Placebos — Placebo will be 5ml vials calculated to equivalent to the 100mg/ml of active drug.
  Arms: Placebo

SUMMARY:
This international, multicentre, pragmatic, double-blind, placebo-controlled, randomised trial of TxA versus placebo will enrol 3,300 patients throughout Australia and internationally. This is an effectiveness trial - some elements of the trial are deliberately left to the perioperative clinicians' discretion in order to reflect usual practice and maximise generalisability.

DETAILED DESCRIPTION:
Study Aims: To conduct a large, multicentre clinical trial of tranexamic acid (TxA), an antifibrinolytic drug routinely used to reduce bleeding in cardiac and some orthopaedic surgery, in 3,300 patients undergoing major gastrointestinal (GI) surgery. Our specific aims are to investigate whether TxA:

Aim 1: Reduces surgical site infection ("wound infection"), and other healthcare-associated infections (pneumonia and sepsis).

Aim 2: Reduces red cell transfusion in GI surgery. Aim 3: Reduces a pooled composite of any serious postoperative complications, and so increases "days alive and at home up to 30 days after surgery" (DAH30).

Aim 4: To evaluate the temporal effect of TxA on perioperative immune and inflammatory responses.

Study Hypothesis Prophylactic TxA administration in patients undergoing major GI surgery reduces the incidence of surgical site infection (SSI) after surgery when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients scheduled for elective or semi-elective (inpatient) open or lap-assisted GI surgery (oesophageal, gastric, hepatobiliary, colorectal) with one or more risk factors for complications:

* Age ≥70 years
* ASA physical status 3 or 4
* Known or suspected history of: heart failure, diabetes, peripheral vascular disease, or chronic respiratory disease
* Obesity (BMI ≥30 kg/m2)
* Anaemia (preoperative haemoglobin <130 g/l in males and <120 g/l in females)
* Renal impairment (se. creatinine ≥150mol/l)
* Low albumin (<30 g/L)

Exclusion Criteria:

* Poor spoken and or written language comprehension
* Laparoscopic cholecystectomy and other minor (eg. closure of stoma) surgery
* Pre-existing infection/sepsis
* Known history of: spontaneous pulmonary embolism, arterial thrombosis familial thrombophilia (e.g. Lupus anticoagulant, protein C deficiency, factor V Leiden)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection | from surgical incision to 30 days post surgical incision
  defined by the US Centers for Disease Control (CDC)

SECONDARY OUTCOMES:
Red cell transfusion | from surgical incision to hospital discharge (from index surgery) or 30 days.
  Total units given
Other healthcare-associated infections | from surgical incision to 30 days
  sepsis, pneumonia, blood stream infection, UTI, etc; all using CDC-guided definitions
C-reactive protein | Postoperative Day 3 (three days after surgical incision)
  peak
Days at home up to 30 days after surgery (DAH30). | From surgical incision to 30 days
  Time that patient spends at home in the 30 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MD, DSc, Study Chair — Alfred Hospital and Monash University
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
This decision will be made on a individual case by case basis, with formal request and review by the PI and steering committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before recruitment of final patient
Access Criteria: Patient and illness eligibility

REFERENCES:
- [Background] O'Higgins N. Endocrine influence on the breast. Ir Med J. 1984 Feb;77(2):49-51. No abstract available. PMID 6538872
- [Background] Takehara K, Nakabayashi Y, Ishibashi Y, Moroi Y, Aikawa T, Inaba K, Meshizuka K. [Immunologic abnormalities in localized scleroderma]. Nihon Hifuka Gakkai Zasshi. 1984 Feb;94(2):121-8. No abstract available. Japanese. PMID 6610780